CLINICAL TRIAL: NCT02078128
Title: To Study the Effect of β-glucans on Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201105013MB
Record Dates: First submitted 2012-09-17; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Burns
Keywords: burn, wound healing, skin graft
MeSH Terms: conditions — Burns | interventions — beta-Glucans; Sugars; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral beta-glucans (Experimental): Daily give kg per day to 30 mg of β-glucan (30mg/kg/day), taking to the wound healed.
  Interventions: Drug: oral sugar powder
- oral sugar powder (Placebo Comparator): control group, daily give and the glucose powder 30 mg per kilogram of body weight (30mg/kg/day) a day, taking to the wound healed.
  Interventions: Dietary Supplement: oral beta-glucans

INTERVENTIONS:
Dietary Supplement: oral beta-glucans — 30 mg/kg, oral every day until wound healed completes or unacceptable toxicity develops.
  Other Names: D-glucose polysaccharides
  Arms: oral sugar powder
Drug: oral sugar powder — 30 mg/kg, oral every day until wound healed completes or unacceptable toxicity develops.
  Other Names: placebo, sugar, glucose
  Arms: oral beta-glucans

SUMMARY:
The purpose of this study is to determine the effect of β-glucans on wound healing.

DETAILED DESCRIPTION:
The structure of βeta-glucan (β-glucans) is a pathogen associated molecular patterns (pathogen-associated molecular patterns, PAMPs), widely present in the cell walls of plants, bacteria, yeasts, fungi, mushrooms and algae. Modern has been reported in the literature that β-glucan can enhance the immune system of animals, and to enhance the function of the animal against bacterial, fungal and viral infections, and cancer.In this study, the use of β-glucan to enhance the biological characteristics of the non-specific immunity, to explore the impact of postoperative patients with wound healing and infection rates.The observation of the healing process to take the Leather District wounds (5 ~ 200 cm2). The experiments were carried out for 18 months, were observed record the following three: (1) the rate of wound healing, (2) The rate of infection assessment: record length of time and the point in time at all levels of antibiotic use also observe the wound change (redness, swelling, heat, pain).(3) days of hospitalization, and spend statistics. Using unpaired student's t-test analysis, group data whether the differences between groups of experimental data. represents a statistically significant when p <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Total burn area under 20%, two to three degree burn and need skin-grafting.
2. Subjects don't have other diseases.
3. Subjects' age between 20 to 60.

Exclusion Criteria:

1. Subjects with hypersensitivity.
2. Subjects with Autoimmune disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Wound healing percentage | every Monday and Thuresday for the duration of hospital stay, an expected average of 3 weeks
  record data by taking picture

CONTACTS AND LOCATIONS:
Overall Officials: Eng Kean Yeong, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan